CLINICAL TRIAL: NCT03228342
Title: The Impact of Musculoskeletal Ultrasound-added to Clinical Evaluations- on Patient Reported Outcomes: A Prospective Study of Rheumatoid Arthritis Patients Classified in Remission/Low Disease Activity (ULTRAPRO)
Brief Title: Ultrasound Impact in Rheumatoid Arthritis Patient Reported Outcomes
Acronym: ULTRAPRO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Clínica de Artritis Temprana (Other)
Collaborators: Instituto Nacional de Ciencias Medicas y Nutricion Salvador Zubiran (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: IRE-2218-17/19-1
Record Dates: First submitted 2017-05-03; First posted 2017-07-24 (Actual); Last update posted 2019-01-30 (Actual); Status verified 2019-01

CONDITIONS: Rheumatoid Arthritis; Patient Reported Outcomes; Musculoskeletal Ultrasound
Keywords: Rheumatoid Arthritis; Ultrasound; Impact
MeSH Terms: conditions — Arthritis, Rheumatoid; Tooth, Impacted

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ultrasound shared (Experimental): Patient will be assessed with ultrasound (GUS-7 score)
  Interventions: Diagnostic Test: MusculoSkeletal Ultrasound
- Ultrasound not shared (Experimental): Patient will be assessed with ultrasound (GUS-7 score)
  Interventions: Diagnostic Test: MusculoSkeletal Ultrasound

INTERVENTIONS:
Diagnostic Test: MusculoSkeletal Ultrasound — Patient will be assess with ultrasound (GUS-7 score) and the results will be informed to his/her attending Rheumatologist.
  The Patient Reported Outcomes will be evaluated a 0,6 and 12 months after randomization.
  Arms: Ultrasound shared
Diagnostic Test: MusculoSkeletal Ultrasound — Patient will be assess with ultrasound (GUS-7 score) and the results will not be informed to his/her attending Rheumatologist.
  The Patient Reported Outcomes will be evaluated a 0,6 and 12 months after randomization.
  Arms: Ultrasound not shared

SUMMARY:
Evaluate the impact of MusculoSkeletal Ultrasound added to Rheumatoid Arthritis patients classified in remission/low disease activity in terms of Patient Reported Outcomes.

ELIGIBILITY:
Inclusion Criteria:

* A clinical diagnosis of RA made at the discretion of the attending experienced rheumatologist.
* Patients classified in remission/low disease activity

Exclusion Criteria:

* <16 years old.
* Patient with recent trauma in the evaluated joints.
* Luxation in the MCP, PIP or MTP joints.

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 94 (Actual)
Dates: Start 2017-05-03 (Actual); Primary Completion 2019-01-28 (Actual); Study Completion 2019-01-28 (Actual)

PRIMARY OUTCOMES:
Change from Baseline of the Patient Reported Outcome (HAQ) | From baseline at 6 months
  Minimal Clinically Significant change in HAQ
Change from Baseline of the Patient Reported Outcome (RADAI) | from baseline at 6 months
  Minimal Clinically Significant change in RADAI
Change from Baseline of the Patient Reported Outcome (SF-36) | from baseline at 6 months
  Minimal Clinically Significant change in SF-36
Change from Baseline of the Patient Reported Outcome (VAS-Patient) | from baseline at 6 months
  Minimal Clinically Significant change in VAS-Patient

SECONDARY OUTCOMES:
Ultrasound findings in Rheumatoid Arthritis Patients Classified in Remission/Low Disease Activity | Baseline
  Describe ultrasound findings at the moment of inclusion in the study.
Clinical relapse: Proportion of patients with relapse after the intervention in both groups | baseline and 6 months
  Describe the proportion of patients with relapse after the intervention in both groups.
Change from Baseline of the Patient Reported Outcome (HAQ) | from baseline at 12 months
  Minimal Clinically Significant change in HAQ
Change from Baseline of the Patient Reported Outcome (RADAI) | from baseline at 12 months
  Minimal Clinically Significant change in RADAI
Change from Baseline of the Patient Reported Outcome (SF-36) | from baseline at 12 months
  Minimal Clinically Significant change in SF-36
Change from Baseline of the Patient Reported Outcome (VAS-Patient) | from baseline at 12 months
  Minimal Clinically Significant change in VAS-Patient

CONTACTS AND LOCATIONS:
Overall Officials: Virginia Pascual, MD, Study Director — INCMNSZ
Locations (1):
- Instituto Nacional de Ciencias Médicas y Nutrición Salvador Zubirán, Mexico City, Mexico

REFERENCES:
- [Background] Plaza M, Nowakowska-Plaza A, Pracon G, Sudol-Szopinska I. Role of ultrasonography in the diagnosis of rheumatic diseases in light of ACR/EULAR guidelines. J Ultrason. 2016 Mar;16(64):55-64. doi: 10.15557/JoU.2016.0006. Epub 2016 Mar 29. PMID 27104003
- [Background] Wakefield RJ, Gibbon WW, Conaghan PG, O'Connor P, McGonagle D, Pease C, Green MJ, Veale DJ, Isaacs JD, Emery P. The value of sonography in the detection of bone erosions in patients with rheumatoid arthritis: a comparison with conventional radiography. Arthritis Rheum. 2000 Dec;43(12):2762-70. doi: 10.1002/1529-0131(200012)43:123.0.CO;2-#. PMID 11145034
- [Background] Nakagomi D, Ikeda K, Okubo A, Iwamoto T, Sanayama Y, Takahashi K, Yamagata M, Takatori H, Suzuki K, Takabayashi K, Nakajima H. Ultrasound can improve the accuracy of the 2010 American College of Rheumatology/European League against rheumatism classification criteria for rheumatoid arthritis to predict the requirement for methotrexate treatment. Arthritis Rheum. 2013 Apr;65(4):890-8. doi: 10.1002/art.37848. PMID 23334942
- [Background] Terslev L, von der Recke P, Torp-Pedersen S, Koenig MJ, Bliddal H. Diagnostic sensitivity and specificity of Doppler ultrasound in rheumatoid arthritis. J Rheumatol. 2008 Jan;35(1):49-53. Epub 2007 Dec 15. PMID 18172922
- [Background] Peluso G, Michelutti A, Bosello S, Gremese E, Tolusso B, Ferraccioli G. Clinical and ultrasonographic remission determines different chances of relapse in early and long standing rheumatoid arthritis. Ann Rheum Dis. 2011 Jan;70(1):172-5. doi: 10.1136/ard.2010.129924. Epub 2010 Nov 19. PMID 21097799
- [Background] Dale J, Purves D, McConnachie A, McInnes I, Porter D. Tightening up? Impact of musculoskeletal ultrasound disease activity assessment on early rheumatoid arthritis patients treated using a treat to target strategy. Arthritis Care Res (Hoboken). 2014 Jan;66(1):19-26. doi: 10.1002/acr.22218. PMID 24376248
- [Background] Smolen JS, Breedveld FC, Burmester GR, Bykerk V, Dougados M, Emery P, Kvien TK, Navarro-Compan MV, Oliver S, Schoels M, Scholte-Voshaar M, Stamm T, Stoffer M, Takeuchi T, Aletaha D, Andreu JL, Aringer M, Bergman M, Betteridge N, Bijlsma H, Burkhardt H, Cardiel M, Combe B, Durez P, Fonseca JE, Gibofsky A, Gomez-Reino JJ, Graninger W, Hannonen P, Haraoui B, Kouloumas M, Landewe R, Martin-Mola E, Nash P, Ostergaard M, Ostor A, Richards P, Sokka-Isler T, Thorne C, Tzioufas AG, van Vollenhoven R, de Wit M, van der Heijde D. Treating rheumatoid arthritis to target: 2014 update of the recommendations of an international task force. Ann Rheum Dis. 2016 Jan;75(1):3-15. doi: 10.1136/annrheumdis-2015-207524. Epub 2015 May 12. PMID 25969430
- [Background] Galicia-Hernandez G, Parra-Salcedo F, Ugarte-Martinez P, Contreras-Yanez I, Ponce-de-Leon A, Pascual-Ramos V. Sustained moderate-to-high disease activity and higher Charlson score are predictors of incidental serious infection events in RA patients treated with conventional disease-modifying anti-rheumatic drugs: a cohort study in the treat-to-target era. Clin Exp Rheumatol. 2016 Mar-Apr;34(2):261-9. Epub 2016 Mar 3. PMID 26939612
- [Background] Backhaus M, Ohrndorf S, Kellner H, Strunk J, Backhaus TM, Hartung W, Sattler H, Albrecht K, Kaufmann J, Becker K, Sorensen H, Meier L, Burmester GR, Schmidt WA. Evaluation of a novel 7-joint ultrasound score in daily rheumatologic practice: a pilot project. Arthritis Rheum. 2009 Sep 15;61(9):1194-201. doi: 10.1002/art.24646. PMID 19714611
- [Background] Backhaus TM, Ohrndorf S, Kellner H, Strunk J, Hartung W, Sattler H, Iking-Konert C, Burmester GR, Schmidt WA, Backhaus M. The US7 score is sensitive to change in a large cohort of patients with rheumatoid arthritis over 12 months of therapy. Ann Rheum Dis. 2013 Jul;72(7):1163-9. doi: 10.1136/annrheumdis-2012-201397. Epub 2012 Sep 6. PMID 22956596
- [Background] Scire CA, Montecucco C, Codullo V, Epis O, Todoerti M, Caporali R. Ultrasonographic evaluation of joint involvement in early rheumatoid arthritis in clinical remission: power Doppler signal predicts short-term relapse. Rheumatology (Oxford). 2009 Sep;48(9):1092-7. doi: 10.1093/rheumatology/kep171. Epub 2009 Jun 26. PMID 19561156
- [Background] Saleem B, Brown AK, Quinn M, Karim Z, Hensor EM, Conaghan P, Peterfy C, Wakefield RJ, Emery P. Can flare be predicted in DMARD treated RA patients in remission, and is it important? A cohort study. Ann Rheum Dis. 2012 Aug;71(8):1316-21. doi: 10.1136/annrheumdis-2011-200548. Epub 2012 Jan 31. PMID 22294638
- [Background] Brown AK, Conaghan PG, Karim Z, Quinn MA, Ikeda K, Peterfy CG, Hensor E, Wakefield RJ, O'Connor PJ, Emery P. An explanation for the apparent dissociation between clinical remission and continued structural deterioration in rheumatoid arthritis. Arthritis Rheum. 2008 Oct;58(10):2958-67. doi: 10.1002/art.23945. PMID 18821687
- [Background] Singh JA, Saag KG, Bridges SL Jr, Akl EA, Bannuru RR, Sullivan MC, Vaysbrot E, McNaughton C, Osani M, Shmerling RH, Curtis JR, Furst DE, Parks D, Kavanaugh A, O'Dell J, King C, Leong A, Matteson EL, Schousboe JT, Drevlow B, Ginsberg S, Grober J, St Clair EW, Tindall E, Miller AS, McAlindon T. 2015 American College of Rheumatology Guideline for the Treatment of Rheumatoid Arthritis. Arthritis Rheumatol. 2016 Jan;68(1):1-26. doi: 10.1002/art.39480. Epub 2015 Nov 6. PMID 26545940
- [Background] Fransen J, Langenegger T, Michel BA, Stucki G. Feasibility and validity of the RADAI, a self-administered rheumatoid arthritis disease activity index. Rheumatology (Oxford). 2000 Mar;39(3):321-7. doi: 10.1093/rheumatology/39.3.321. PMID 10788543
- [Background] El Miedany Y, El Gaafary M, Palmer D. Assessment of the utility of visual feedback in the treatment of early rheumatoid arthritis patients: a pilot study. Rheumatol Int. 2012 Oct;32(10):3061-8. doi: 10.1007/s00296-011-2098-1. Epub 2011 Sep 11. PMID 21909946
- [Background] Wolfe F, Pincus T. Listening to the patient: a practical guide to self-report questionnaires in clinical care. Arthritis Rheum. 1999 Sep;42(9):1797-808. doi: 10.1002/1529-0131(199909)42:93.0.CO;2-Q. No abstract available. PMID 10513792
- [Background] Kosinski M, Zhao SZ, Dedhiya S, Osterhaus JT, Ware JE Jr. Determining minimally important changes in generic and disease-specific health-related quality of life questionnaires in clinical trials of rheumatoid arthritis. Arthritis Rheum. 2000 Jul;43(7):1478-87. doi: 10.1002/1529-0131(200007)43:73.0.CO;2-M. PMID 10902749
- [Background] Anderson JK, Zimmerman L, Caplan L, Michaud K. Measures of rheumatoid arthritis disease activity: Patient (PtGA) and Provider (PrGA) Global Assessment of Disease Activity, Disease Activity Score (DAS) and Disease Activity Score with 28-Joint Counts (DAS28), Simplified Disease Activity Index (SDAI), Clinical Disease Activity Index (CDAI), Patient Activity Score (PAS) and Patient Activity Score-II (PASII), Routine Assessment of Patient Index Data (RAPID), Rheumatoid Arthritis Disease Activity Index (RADAI) and Rheumatoid Arthritis Disease Activity Index-5 (RADAI-5), Chronic Arthritis Systemic Index (CASI), Patient-Based Disease Activity Score With ESR (PDAS1) and Patient-Based Disease Activity Score without ESR (PDAS2), and Mean Overall Index for Rheumatoid Arthritis (MOI-RA). Arthritis Care Res (Hoboken). 2011 Nov;63 Suppl 11:S14-36. doi: 10.1002/acr.20621. No abstract available. PMID 22588741
- [Background] Lillegraven S, Prince FH, Shadick NA, Bykerk VP, Lu B, Frits ML, Iannaccone CK, Kvien TK, Haavardsholm EA, Weinblatt ME, Solomon DH. Remission and radiographic outcome in rheumatoid arthritis: application of the 2011 ACR/EULAR remission criteria in an observational cohort. Ann Rheum Dis. 2012 May;71(5):681-6. doi: 10.1136/ard.2011.154625. Epub 2011 Oct 12. PMID 21994234
- [Background] Fransen J, van Riel PL. Outcome measures in inflammatory rheumatic diseases. Arthritis Res Ther. 2009;11(5):244. doi: 10.1186/ar2745. Epub 2009 Oct 14. PMID 19849821